CLINICAL TRIAL: NCT02057068
Title: Improving Sleep In Veterans and Their Family Caregivers
Brief Title: Improving Sleep in Veterans and Their CGs
Acronym: SLEEP-E Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: E7249-W
Record Dates: First submitted 2014-01-24; First posted 2014-02-06 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Sleep Quality
Keywords: Caregivers; Telemedicine; Sleep Disorders; Meditation; Cognitive Behavioral Therapy; Activity Enhancement; Technology; Non-pharmacological sleep intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Randomization to an immediate intervention group or a no-contact wait list control group. Following post intervention assessments the wait-list control group received the intervention.
Masking Description: This efficacy study was not blinded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLEEP-E Dyads Intervention (Experimental): SLEEP-E Dyads Six-Week Tele-Health Intervention
  1. . Daily core video modules on sleep education, sleep hygiene and behavioral and environmental factors influencing sleep.
  2. . Daily and on-demand video modules designed to promote and provide guided instruction for daily "Move Out" time consisting of activity enhancement and exercise.
  3. . Daily and on-demand video modules designed to promote and provide guided instruction for daily "Stand Down" time (meditation, therapeutic breathing and self-care).
  4. . SLEEP-E Dyads book
  5. . Two tele-video conferences to discuss evaluation results, obtain buy-in for the prescribed intervention and address dysfunctional beliefs and attitudes about sleep. The second call involves checking-in, encouragement, reinforcement and coaching
  Interventions: Behavioral: SLEEP-E Dyads Intervention
- Usual Care Group (No Intervention): During the intervention period there is no data collection or contact with research staff other than for scheduling outcomes visits.

INTERVENTIONS:
Behavioral: SLEEP-E Dyads Intervention — Described in arm/group description
  Arms: SLEEP-E Dyads Intervention

SUMMARY:
This study addresses the neglected topic of sleep disturbance in older caregiving dyads-a topic that has important implications for the safety, health, functioning and quality of life of older Veterans living at home and being cared for by a family caregiver (CG). The purpose of the study was to develop and field test non-pharmacological, technology enhanced sleep hygiene, exercise and meditation interventions to improve sleep in Veteran caregiving dyads.The conceptual framework of the intervention incorporated components of cognitive behavioral therapy, psycho-education and self-management support for individuals with chronic conditions with an emphasis on cultivating competence and mastery.

DETAILED DESCRIPTION:
Research Plan:

Sample. Veteran care receivers(CR s) or carepartners (CP) over the age of 60 who require assistance from a spousal or cohabitating caregiver (CG) and Veteran caregivers providing care for a cohabitating carepartner were recruited. Dyads underwent comprehensive baseline assessments consisting of in-person home-based interviews and iPad training (T1) followed by a week-long data collection of contemporaneous actigraphic sleep parameters and twice daily (morning and evening) indices of subjective sleep, activity, mood, behavior and sleep hygiene completed on the Tonic for Health Platform. Dyads were randomly assigned to an immediate intervention or wait-list control group. The immediate group received the intervention described below followed by post-intervention assessments (T2) identical to baseline. Wait-list participants then received the intervention followed by a final post-intervention assessment for the wait-list group only (T3).

Intervention.

Daily Videos: Video modules were delivered daily to the dyads' iPads during the 6-week intervention. All participants received core programming of sleep hygiene education, and guided instruction for daily physical activity enhancement "Move-Out!" and meditation/relaxation/self-care "Stand Down!" sessions individualized to functional ability levels. The baseline data allowed for subsequent compilation and programming of individualized, algorithmically derived, adaptive prescriptions for relevant video modules, sleep hygiene recommendations and cognitive behavioral strategies based upon the three independent streams of objective and subjective data for each dyad member. During the intervention dyads completed brief morning and evening diaries to assess compliance with the intervention and capture daily mood and sleep/sleep hygiene data.

Tele-Video-Conferences: Each dyad participated in two tele-video conferences with the PI. The first was to discuss evaluation results, obtain buy-in for the prescribed intervention and address dysfunctional beliefs and attitudes about sleep. The second call was a check-in, encouragement, reinforcement and coaching call. Dyads were re-assessed following the 6-week intervention.

Evaluations:

Standardized quantitative evaluations regarding the utility of the program were completed following the post-intervention assessments on the iPads. A sub-sample of dyads also participated in qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Care recipient must be age 60 and over and require assistance from the identified caregiver with more than one Activity of Daily Living or three or more Instrumental Activities of Daily Living,
* have a life expectancy of greater than or equal to six (6) months,
* have no plans for transitioning out of home in the next six months,
* and have approval from the primary care provider to participate in the research.
* Caregivers must live with care recipient
* Caregivers must obtain a negative mini-cog assessment or negative TICS-m assessment. Caregivers can be any relation (spouse, child, sibling, friend, etc.) to the care recipient so long as the two are cohabitating.
* Caregiver can be any age.
* For Phase 2 and Phase 3 of the study, either the care recipient or the caregiver must have difficulty sleeping as indicated by scores on the Insomnia Severity Index.

Exclusion Criteria:

* Parkinson's with tremor or other movement disorder that would invalidate actigraphy
* Untreated diagnosis of sleep apnea or restless leg syndrome
* Inability to tolerate actigraphy
* CG and CR sleep efficiency > 85% and/or both members of dyad report sleeping well
* Caregivers must have a negative screen with the Mini-Cog or the ModifiedTelephone Interview for Cognitive Status (TICS-M) to demonstrate cognitive capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Griffiths, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the intervention occurred between 2014 and 2016. Participants were recruited from the Geriatrics Clinic, the CVNR Caregiver Registry and by referrals from Social Workers and Primary Care.
Pre-assignment Details: Participants were excluded from the study if both members of the dyad reported sleeping well (no sleep problems, high sleep quality) during baseline interview and/or had sleep efficiency of 85% or greater as measured by actigraphy during baseline week. Randomization occurred following baseline. Consented=102; Randomization=96.
Groups:
- SLEEP-E Dyads Intervention: SLEEP-E Dyads Intervention
  Adaptive prescriptions for the individualized components of the sleep intervention will be written for each dyad based upon dyad-specific risk factors, sources of sleep disturbance, nature of sleep problems and baseline sleep hygiene practices. In addition, each dyad will receive a core intervention component consisting of a sleep hygiene psycho-education curriculum, activity enhancement and relaxation instruction and training delivered by the iPads and two tele-video conferences to discuss evaluation, obtain buy-in for the intervention and provide coaching.
- Wait List Control Group: During the intervention period there is no data collection or contact with research staff other than for scheduling outcomes visits.
Period: Overall Study
Arm/Group | SLEEP-E Dyads Intervention | Wait List Control Group
Started (12 beta test dyads included in the intervention group, thus they were not randomized.) | 60 | 36
Completed | 52 | 28
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Caregiver (CG) Health | 0 | 2
Not completed — Carepartner (CP) Health | 4 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Dyads completed a comprehensive interview followed by a weeklong in-home sleep assessment (actigraphy) and journals. Dyads who didn't complete the week were excluded. Others reported sleeping well and were excluded based on that and/or actigraphic assessments. Dyads were randomized after baseline. Only completers were enrolled.
Groups:
- SLEEP-E Dyads Intervention: SLEEP-E Dyads Six-Week Tele-Health Intervention
  1. . Daily core video modules on sleep education, sleep hygiene and behavioral and environmental factors influencing sleep.
  2. . Daily and on-demand video modules designed to promote and provide guided instruction for daily "Move Out" time consisting of activity enhancement and exercise.
  3. . Daily and on-demand video modules designed to promote and provide guided instruction for daily "Stand Down" time (meditation, therapeutic breathing and self-care).
  4. . SLEEP-E Dyads book
  5. . Two tele-video conferences to discuss evaluation results, obtain buy-in for the prescribed intervention and address dysfunctional beliefs and attitudes about sleep. The second call involves checking-in, encouragement, reinforcement and coaching
  SLEEP-E Dyads Intervention: Described in arm/group description
- Total: Total of all reporting groups
Arm/Group | SLEEP-E Dyads Intervention | Usual Care Group | Total
Number analyzed (Participants) | 60 | 36 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline measures were collected in the home of the dyads by trained interviewers.
  In addition dyads completed morning and evening daily diaries for 7 days.
  Years | 70.12 (8.14) | 70.11 (9.43) | 70.12 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This was dyadic data involving a Veteran and a co-habitating caregiver or a Veteran caregiver and his/her care-partner
  Participants
    Female | 30 | 18 | 48
    Male | 30 | 18 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 36 | 96

OUTCOME MEASURES:

1. Primary Outcome: Subjective Sleep Quality
Description: Pittsburgh Sleep Quality Index Scores (PSQI) The Pittsburgh Sleep Quality Index is a standardized and validated measure of subjective sleep quality and sleep disturbance. The inventory has 18-items. PSQI scores range from 0 - 21. A total score > 5 (some evidence for 8) is indicative of poor sleep quality.
Time Frame: Baseline (T1) and Post-Intervention (T2) - 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SLEEP-E Dyads Intervention | Wait List Control Group
Number analyzed (Participants) | 60 | 36
units on a scale
  Baseline | 8.41 (3.64) | 8.31 (4.03)
  Post Intervention | 5.98 (2.84) | 8.63 (4.19)
Statistical Analysis 1: Comparison: SLEEP-E Dyads Intervention vs Wait List Control Group; Test type: Superiority; p < .001, ANOVA; Intention to treat analysis with last observation carried forward; Partial Eta Squared = .282

2. Secondary Outcome: Mean Sleep Efficiency
Description: Average sleep efficiency over 7 nights of actigraphic measurement . Sleep efficiency is calculated as the number of hours asleep divided by the number of hours in bed with the intention to sleep.
Time Frame: Baseline (T1) and Post-Intervention (T2) - 8 Weeks
Measure: Mean (Standard Deviation); unit: percentage of sleep/time in bed
Arm/Group | SLEEP-E Dyads Intervention | Usual Care Group
Number analyzed (Participants) | 60 | 36
percentage of sleep/time in bed
  Baseline | 82.19 (6.71) | 82.55 (5.71)
  Post Intervention | 81.64 (7.26) | 82.09 (6.11)
Statistical Analysis 1: Comparison: SLEEP-E Dyads Intervention vs Usual Care Group; Test type: Superiority — Intention to treat analysis with last observation carried forward; p > .05, ANOVA

3. Secondary Outcome: BEF-SHI Total Number of Negative Sleep Hygiene Behaviors
Description: Total Number of negative sleep hygiene indicators from the BEFSHI - Bedtime Environmental Features and Sleep Hygiene Index (e.g., nighttime caffeine, nighttime snacking-sugar, nicotine, excessive alcohol, excessive daytime napping, television, tablet and computer use in bedroom after 9 pm etc.) Participants are asked to respond yes (1) or no (0) to a series of sleep hygiene behaviors considered detrimental to sleep. Scores are summed. Possible scores range from 0-8 with a greater score indicating a greater number of negative sleep hygiene behaviors endorsed.
Time Frame: Baseline (T1) and Post-Intervention (T2) - 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SLEEP-E Dyads Intervention | Usual Care Group
Number analyzed (Participants) | 60 | 36
units on a scale
  Baseline | 5.27 (2.21) | 4.39 (2.27)
  Post Intervention | 3.12 (2.08) | 4.51 (2.12)
Statistical Analysis 1: Comparison: SLEEP-E Dyads Intervention vs Usual Care Group; Test type: Superiority; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: Data were collected throughout the study. There were no adverse events.
Groups:
- SLEEP-E Dyads Intervention: SLEEP-E Dyads Intervention
  Adaptive prescriptions for the individualized components of the sleep intervention will be written for each dyad based upon dyad-specific risk factors, sources of sleep disturbance, nature of sleep problems and baseline sleep hygiene practices. In addition, each dyad will receive a core intervention component consisting of a sleep hygiene psycho-education curriculum, activity enhancement and relaxation instruction and training delivered by the iPads and two tele-video conferences to discuss evaluation, obtain buy-in for the intervention and provide coaching.
  There were no adverse events.
- Wait List Control Group: During the intervention period there is no data collection or contact with research staff other than for scheduling outcomes visits. There were no adverse events.
Arm/Group | SLEEP-E Dyads Intervention | Wait List Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/36
Other Adverse Events (participants affected / at risk) | 0/60 | 0/36

LIMITATIONS AND CAVEATS:
This was a pilot and feasibility study involving dyads who self-selected into the program. The sample size is small, thus the results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No